CLINICAL TRIAL: NCT05115695
Title: The Effect of Different Upper Extremity Strengthening Trainings on Functionality, Muscle Strength and Trunk in Children With Cerebral Palsy in Kahramanmaras
Brief Title: The Effect of Upper Extremity Strengthening on Functionality, Muscle Strength and Trunk in Children With Cerebral Palsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kahramanmaras Sutcu Imam University (Other)
Responsible Party: Principal Investigator, Hatice Adiguzel, assistant professor, Kahramanmaras Sutcu Imam University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: hatice
Record Dates: First submitted 2021-10-13; First posted 2021-11-10 (Actual); Last update posted 2023-10-11 (Actual); Status verified 2023-10

CONDITIONS: Cerebral Palsy; Upper Extremity Dysfunction; Upper Extremity Functions; Muscle Strength; Cerebral Palsy, Spastic; Cerebral Palsy Spastic Diplegia
Keywords: Cerebral Palsy; Upper Extremity Dysfunction; Upper Extremity Strengthening; muscle strength; trunk; functionality; Proprioceptive Neuromuscular Facilitation
MeSH Terms: conditions — Cerebral Palsy | interventions — Muscle Stretching Exercises

STUDY DESIGN:
Intervention Model Description: The study will include 30 children with cerebral palsy (CP) diagnosed at the GMFCS I-II level with 15 controls and 15 treatment groups. Included individuals (n=30) will be randomized by simple random method and divided into 2 groups. 2 groups; different upper extremity strengthening training and 1 grup (n=15,control): Neurodevelopmental Treatment (NDT-Bobath) approaches will be applied to the second group for 6 weeks, 3 days a week, 45 minutes a day. Group 2: An exercise approach with Proprioceptive Neuromuscular Facilitation (PNF) (n=15, exercise group) UE patterns will be applied to the first group for 30 minutes, 3 days a week for 6 weeks.
Who Masked: Outcomes Assessor
Masking Description: Evaluations will be made twice, before and after the treatment. All assessments will be made by a different physician physiotherapist who is unfamiliar with the treatment groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PNF/Interventional (Active Comparator): Upper extremity and scapular patern of PNF exercise approach will be applied to the first group for 6 weeks, 3 days a week, 30 minutes a day.
  Interventions: Other: muscle strengthening exercise/Proprioceptive Neuromuscular Facilitation (PNF)
- NDT/Experimental (Experimental): Upper extremity strengthening exercises consisting of Neurodevelopmental Therapy (NGT-Bobath) approaches will be applied to the second group for 45 minutes, 3 days a week for 6 weeks.
  Interventions: Other: traditional physiotherapy approach

INTERVENTIONS:
Other: traditional physiotherapy approach — Traditional upper extremity strengthening and tonus regulation (weight shifting, weight bearing, active reaching in sitting exercises) exercises consisting of Neurodevelopmental Therapy (NDT-Bobath) approaches will be applied to the second group for 45 minutes, 3 days a week for 6 weeks.
  Other Names: Neurodevelopmental Therapy (NDT-Bobath)
  Arms: NDT/Experimental
Other: muscle strengthening exercise/Proprioceptive Neuromuscular Facilitation (PNF) — Muscle strengthening with scapular and upper extremity patterns of PNF exercise approach will be applied to the first group for 6 weeks, 3 days a week, 30 minutes a day.
  Other Names: Proprioceptive Neuromuscular Facilitation (PNF)
  Arms: PNF/Interventional

SUMMARY:
Cerebral Palsy (CP) is an activity limitation, movement and posture deficiencies in early stage of life. In 80% of these children, upper extremity (UE) dysfunctions are observed, which leads to loss of quality of life, resulting in limited participation in activities of daily living (ADL). When the hands are affected in UE, fine motor skills such as grasping, writing and object manipulation are usually limited. This results in inadequate use of the extremities in functional activities. Although all children with CP are known to be affected by UE, studies in terms of physiotherapy and rehabilitation methods mostly focused on children with hemiparetic CP. Similar problems are observed in children with bilateral involvement. However, a wide variation is observed in the bimanual performance of children with hemiparetic and bilateral involvement. Studies evaluating UE activities in children with CP; emphasized that the inability to manipulate objects manually is one of the most important reasons for the restriction of participation in ADLs. Physiotherapy and rehabilitation programs include many neurodevelopmental treatment approaches including stretching, strengthening, positioning, splinting, casting, orthosis selection and movement facilitation. However, it is known that studies investigating the current efficacy of these treatments on UE functions mostly focus on unilateral CP. Interventions that focus on improving UE functions in children with bilateral CP are limited. In UE rehabilitation in bilateral CP; states that target-focused therapy, bimanual intensive task specific training programs and trainings such as HABIT (intensive bimanual training of the upper extremity) involving the lower extremity have been used, but there is only evidence for HABIT-ILE (HABIT involving the lower extremity). In the literature, it is observed that strengthening training with the Proprioceptive Neuromuscular Facilitation (PNF) method, which makes a significant contribution to muscle strength balance, is mostly used in lower extremity rehabilitation in these children. In this study, in the UE rehabilitation of children with hemiparetic and diparetic CP; in order to stimulate motor responses and improve neuromuscular control and function, the superiority of the PNF approach applied with scapular and UE patterns over the traditional Neurodevelopmental Therapy (NGT-Bobath) method will be determined.

DETAILED DESCRIPTION:
European SP Surveillance (SCPE), CP subtypes according to the dominant type of tone and movement abnormality; divided into spastic, dyskinetic and ataxic CP. Spastic type SP; unilateral spastic (hemiparetic) and bilateral (quadriparetic and diparetic), dyskinetic SP; defined as dystonic and choreoathetotic. Spastic type constitutes 90% of this population and bilateral/unilateral involvement is observed in this group. In 80% of these children, upper extremity (UE) dysfunctions are observed, which leads to loss of quality of life, resulting in limited participation in activities of daily living (ADL).Children with CP as a result of damage to the motor cortex and corticospinal tracts; develop abnormal movement patterns by having difficulties in reaching, grasping and fine motor skills of UE. When the hands are affected in UE, fine motor skills such as grasping, writing and object manipulation are usually limited. This results in inadequate use of the extremities in functional activities. Although all children with CP are known to be affected by UE, studies in terms of physiotherapy and rehabilitation methods mostly focused on children with hemiparetic CP. The most common in children with hemiparetic CP; increase in muscle tone and decreased normal joint movement (ROM), decrease in UE muscle and grip strength, primitive grasping reflex, loss of speed and dexterity are observed. In addition to pure motor impairment, sensorimotor problems are also observed. Similar problems are observed in children with bilateral involvement. However, a wide variation is observed in the bimanual performance of children with hemiparetic and bilateral involvement. Studies evaluating UE activities in children with CP; emphasized that the inability to manipulate objects manually is one of the most important reasons for the restriction of participation in ADLs. In a study examining UE disorders, hand dexterity, grip strength and functionality in ADLs in children with diparetic CP; it was emphasized that these children also had deficiencies in dexterity, grip strength and functions in ADL. Therefore, it has been shown that these children are also negatively affected in terms of hand skills, coordination, UE muscle strength, grip strength, ADL and functional skills compared to their healthy peers. Observing that UE rehabilitation in CP remains in the background, studies on the pathophysiology and treatment of UE sequelae in the last 5 years have come to the fore. Physiotherapy and rehabilitation programs; it includes many neurodevelopmental treatment approaches including stretching, strengthening, positioning, splinting, casting, orthosis selection and movement facilitation. However, it is known that studies investigating the current efficacy of these treatments on UE functions mostly focus on unilateral CP. Interventions that focus on improving UE functions in children with bilateral CP are limited. In UE rehabilitation in bilateral CP; states that target-focused therapy, bimanual intensive task specific training programs and trainings such as HABIT (intensive bimanual training of the upper extremity) involving the lower extremity have been used, but there is only evidence for HABIT-ILE (HABIT involving the lower extremity). In the literature, it is observed that strengthening training with the Proprioceptive Neuromuscular Facilitation (PNF) method, which makes a significant contribution to muscle strength balance, is mostly used in lower extremity rehabilitation in CP. In this study, in the UE rehabilitation of children with hemiparetic and diparetic CP; in order to stimulate motor responses and improve neuromuscular control and function, the superiority of the PNF approach applied with scapular and UE patterns over the traditional Neurodevelopmental Therapy (NGT-Bobath) method will be determined. As a result of this study, it is thought that in addition to traditional NGT-Bobath treatment approaches, muscle strengthening with scapular pattern and upper extremity patterns of PNF can be an effective treatment alternative in the UE rehabilitation of children with CP, and it is thought that UE functional skills, muscle strength and trunk control of individuals will be positively affected. Included children will be randomized by simple randomisation and divided into 2 groups. An exercise approach with PNF UE patterns will be applied to the first group for 30 minutes, 3 days a week for 6 weeks. UE rehabilitation consisting of Neurodevelopmental Treatment (NGT-Bobath) approaches will be applied to the second group for 6 weeks, 3 days a week, 45 minutes a day. Treatments will be carried out by the same doctor physiotherapist investigator. Evaluations will be made twice, before and after the treatment. All assessments will be made by a blind doctor physiotherapist investigator who is unfamiliar with the treatment groups. Alongside the studies in the literature, this study will be the first to compare the effectiveness of the use of UE patterns of PNF in children with hemiparetic and diparetic CP.

ELIGIBILITY:
Inclusion Criteria:

1. Having been diagnosed with CP according to SCPE criteria
2. Be between 8-18 years old
3. Volunteering to participate in the study
4. Hand functions 1-2 according to MACS
5. To be at the level of 1-2-3 according to the GMFCS (Gross Motor Function Classification System)
6. Individuals with hemiparetic-diparetic CP who can take verbal commands
7. Upper extremity muscle tone ≤ 2 according to Modified Ashworth Scale (MASH)

Exclusion Criteria:

1. Less than 8 years old, over 18 years old
2. Receiving any UE surgery / Botulinum toxin (Btx) treatment in the last 6 months
3. Having other known neurological disease
4. Any upper extremity contracture

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2023-01-15 (Actual); Study Completion 2023-01-30 (Actual)

PRIMARY OUTCOMES:
The change of Manual Ability Classification System (MACS) | first day of intervention and after the 6 weeks
  Manual Ability Classification System will be used in hand skills for the evaluation of upper extremity. MACS is a system that classifies children's ability to handle objects during their daily activities. While MACS evaluates the participation of both hands in activities together, it does not evaluate the hands separately.
The change of the Abilhand Kids Scale | first day of intervention and after the 6 weeks
  The Abilhand Kids scale is the Abilhands Kids questionnaire, a parent questionnaire that describes the child's ease or difficulty in performing bilateral activities for the assessment of upper extremity skills. 21 items; relates to activities of daily living, such as taking off a T-shirt, filling a glass of water, or putting on a backpack. Scoring items; recorded as impossible, difficult, or easy. After the survey is completed, it is scored regardless of how the items are completed. A maximum total of 42 points is obtained. Scores are '0 = Impossible', '1 = Difficult' and '2 = Easy'. A maximum of 42 points can be obtained. Higher score indicates better score.
The change of the Jebsen-Taylor Hand Function Test (JEFT) | first day of intervention and after the 6 weeks
  The Jebsen-Taylor Hand Function Test (JEFT) consists of a series of subtests representing hand functions in daily life for the evaluation of hand functions. Separate tests are performed for the dominant and non-dominant extremities, and the time to perform five tests for each hand is recorded in seconds. Apart from the sub-parameter of writing, a total of 6 functions, including turning the page, throwing small objects into the box, warning to eat, lining up the checkerboards, lifting large-light objects and lifting large-heavy objects, are standardized and implemented.
The change of the 9-hole Peg test (9DPT) | first day of intervention and after the 6 weeks
  The 9-hole Peg test (9DPT) is one of the most commonly used tools to assess dexterity. It is an upper extremity skill test that can be completed in a short time. Tests can be done on both hands. Test materials consist of nine holes on a flat, small test battery and nine wooden sticks that fit into them. The subjects are asked to take the rods one by one from the chamber at the top of the test battery and place them in the holes at the bottom of the chamber without any order, then take the rods out of the holes and put them in the upper chamber. Time taken to complete the test, sec. recorded in . The test is reliable and valid.
The change of the Purdue-Peg board test | first day of intervention and after the 6 weeks
  The Purdue-Peg board test (PPBT) is one of the most commonly used tests for selecting personnel for jobs that require motor skills and coordination. It is a test that also measures fingertip dexterity required in assembly works. Washers, rings and small nails are used in this test. The test completion time is recorded in seconds. The test is valid and reliable.
The change of the strength of upper extremity muscle | first day of intervention and after the 6 weeks
  Strength of bilateral pectorals, rhomboids, serratus anterior, trapezius, deltoid, supraspinatus, infraspinatus, teres minor, biceps brachy, wrist extensors and flexors with digital muscle strength measurement device ((Commander Echo Base Kit+Echo Muscle Tester (J-Tech)).
The change of the Trunk Control Measurement Scale (TCMS) | first day of intervention and after the 6 weeks
  The Trunk Control Measurement Scale (TCMS) consists of two main parts: static sitting balance and dynamic sitting balance. Static sitting balance examines static trunk control during movements of the upper and lower extremities. Dynamic control of sitting; It is divided into two as selective motor control and dynamic reach. Selective control of dynamic sitting balance is a scale that evaluates certain movements of the trunk in three planes (flexion, extension, lateral flexion and rotation). Total score ranges between 0 and 58 and higher scores reflect better control.
Hand grip strength | first day of intervention and after the 6 weeks
  Hand grip strength will be measured with Jamar hand dynamometer.
Pinch grip strength | first day of intervention and after the 6 weeks
  Pinch grasp strength will be measured by Pinch Meter.

SECONDARY OUTCOMES:
The change of the Modified Ashworth Scale (MASH) | first day of intervention and after the 6 weeks
  The Modified Ashworth Scale (MASH) is a method used to determine the severity of spasticity. It is based on the subjective rating of the resistance felt during the examination. Spasticity of the bilateral pectoralis, elbow flexors, pronators, wrist and finger flexors muscles in the upper extremity will be evaluated. The tone felt in these muscles against passive movement is classified as follows; 0: No increase in tone, 1: Slight increase in tone characterized by catching and relaxation or mild resistance at the end of the ROM, 1+: Slight increase in tone characterized by minimal resistance in the remaining ROM (less than half) after capture, 2: Significant tone over most of the ROM increase, but the affected joint can be moved easily, 3: Significant increase in muscle tone, passive movement is difficult, 4: The involved part is rigid in flexion or extension.

CONTACTS AND LOCATIONS:
Overall Officials: zekiye ipek katirci kirmaci, PhD, Study Chair — Kahramanmaras Sutcu Imam University; mehmet göğremiş, PhD, Study Chair — Kahramanmaras Sutcu Imam University; Deniz Tuncel Berktas, Proffessor, Study Chair — Kahramanmaras Sutcu Imam University; Cengiz Dilber, Proffessor, Study Chair — Kahramanmaras Sutcu Imam University
Locations (1):
- Kahramanmaras Sutcu Imam University, Kahramanmaraş, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No